CLINICAL TRIAL: NCT03245203
Title: A Pilot Study of Neoadjuvant Chemotherapy Combined With Bevacizumab for Locally Advanced Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, DuNan, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170801001
Record Dates: First submitted 2017-08-01; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Rectal Cancer
Keywords: neoadjuvant chemotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 70 patients with rectal adenocarcinoma clinical staging in Stage II or Stage III were included for neoadjuvant therapy followed by TME, of which 35 underwent neoadjuvant radiotherapy, and other 35 underwent neoadjuvant chemotherapy+beacizumab.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): beacizumab+ neoadjuvant chemotherapy (FOLFIRI+beacizumab)
  Interventions: Procedure: FOLFIRI+beacizumab
- Control group (Active Comparator): neoadjuvant CRT for consecutive 5 weeks
  Interventions: Procedure: CRT

INTERVENTIONS:
Procedure: FOLFIRI+beacizumab — Eligible patients received bevacizumab 5.0 mg/kg followed by irinotecan 125mg/m2 combined with LV 200mg/m2 followed by 5-FU bolus 400mg/m2,then 5-FU infusion 2.4~3.0g/m2 over a 46-h period.Those agents were given for a 2-week cycle.Treatment was administered for six cycles. LARC was reevaluated and operated after 4~8 weeks.
  Arms: Experimental group
Procedure: CRT — total dose of radiotherapy was 40~50Gy, a subdose of 1.8~2Gy for continuous 5 weeks, 5 times/week.Then,5-FU infusion 400mg/m2 combined with LV 200mg/m2 over 24 h for 4 days/week during the first and fifth weeks of radiotherapy.Whereas,Capecitabine was administered orally at a dose of 825mg/m2 twice a day for 5 days of a week. Second staging and operation were performed in the sixth week after chemoradiotherapy.
  Arms: Control group

SUMMARY:
Background: Neoadjuvant chemoradiotherapy (CRT) and total mesorectum excision (TME) has become the standard therapy for the treatment of locally advanced rectal cancer (LARC) to reduce the local recurrence rate, however, no improvement of distant metastasis rate was observed, and the incidence of postoperative local recurrence and distant metastasis can reach more than 25%. It is still a challenge for us to improve the RO resection rate of locally advanced rectal cancer and reduce the incidence of local recurrence and distant metastasis.

DETAILED DESCRIPTION:
Objective: compared with the postoperative adjuvant therapy, neoadjuvant chemotherapy has shown better compliance of LARC patients, and may be more effective in reducing the incidence of local recurrence and distant metastasis. This study used the anti-angiogenesis drugs beacizumab and chemotherapy in patients with LARC for neoadjuvant chemotherapy, and investigated the short-term efficacy to provide objective basis for the selection of neoadjuvant therapy.

Methods: 70 patients with rectal adenocarcinoma clinical staging in Stage II or Stage III were included for neoadjuvant therapy followed by TME, of which 35 underwent neoadjuvant radiotherapy, and other 35 underwent neoadjuvant chemotherapy+beacizumab.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical stage II or stage III rectal cancer patients diagnosed by preoperative biopsy pathology report, endoscopic examination report and preoperative abdominal pelvic dynamic contrast enhanced-MRI examination (DCE-MRI); 2. Primary tumor lesions within 4~12 cm from the anus through endoscopic examination; 3. No distant metastasis and intestinal obstruction; 4. No surgical contraindications; 5. Can be treated with neoadjuvant chemotherapy confirmed by normal routine examination; 6. informed consent with patients and family members before treatment.

Exclusion Criteria:

* history of beacizumab allergy, being treated with other therapy important viscera dysfunction and severe heart disease, including congestive heart failure, arrhythmia beyond the control, long-term drug treatment of angina pectoris, heart valve disease, myocardial infarction, and resistant hypertension; infectious wound and uncontrollable history of mental illness; infectious sexual diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3 years
  percent

SECONDARY OUTCOMES:
disease-free survival (DFS) | 3 years
  year
overall survival (OS) | 3 years
  year
overall response rate (ORR) | 3 years
  percent

CONTACTS AND LOCATIONS:
Overall Officials: nan du, Principal Investigator — First Affiliated Hospital, Chinese PLA General Hospital
Locations (1):
- First Affiliated Hospital, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No